CLINICAL TRIAL: NCT03835741
Title: Reduction of Length of Stay by Automated Adjustment of Oxygen on Patient With Acute COPD Exacerbation - FreeO2 HypHop
Brief Title: Automated Adjustment of Oxygen on Patient With Acute COPD Exacerbation - FreeO2 HypHop
Acronym: FreeO2 HypHop
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The clinical implementation of the system used in the study as well as its routine use limited the possibilities of carrying out this project.
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, François Lellouche, Principal Investigator, Laval University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21641
Record Dates: First submitted 2019-01-14; First posted 2019-02-11 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Oxygen Toxicity; COPD Exacerbation; Hyperoxia; Hypoxemia; Hypoxic Respiratory Failure
MeSH Terms: conditions — Hyperoxia; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Automated Oxygen titration (Experimental): In this arm, an automated adjustment of oxygen during patient hospitalisation by FreeO2 device
  Interventions: Device: FreeO2
- Manual Oxygen titration (Other): In this arm, a manual adjustment of oxygen during patient hospitalisation by hospital staff
  Interventions: Other: manual titration

INTERVENTIONS:
Device: FreeO2 — an automated adjustment of oxygen during patient hospitalisation by FreeO2 device
  Arms: Automated Oxygen titration
Other: manual titration — a manual adjustment of oxygen during patient hospitalisation by hospital staff
  Arms: Manual Oxygen titration

SUMMARY:
The aim of this study is to evaluate if automated adjustment of oxygen (with FreeO2 device) can reduce the hospital length of stay for acute exacerbation of COPD with comparison of manual oxygen titration.

DETAILED DESCRIPTION:
The aim of this study is to evaluate if automated adjustment of oxygen (with FreeO2 device) can reduce the hospital length of stay for acute exacerbation of COPD with comparison of manual oxygen titration.

Patients with severe acute exacerbation of COPD requiring hospitalization will be included in this randomized controlled study and will be managed with either manual oxygen titration or automated oxygen titration (FreeO2 arm).

The impact on the hospital length of stay will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* COPD or suspected COPD ( Age>40, active or smoking history > 10pack/years), -
* Acute exacerbation (increasing dyspnea recently)
* One or more of the following criteria: increased sputum, modification of sputum purulence,increased dyspnea,
* Moderate oxygen therapy: Oxygen flow < 8 lpm (or FiO2 < 0.60) to maintain a SpO2 >or = 92% (for long term oxygen therapy, the oxygen flow must be greater than baseline flow to maintain SpO2 > or = 92%)

Exclusion Criteria:

* Patient refusal
* COPD exacerbation with diagnosis highly related to pulmonary embolism, cardiac pulmonary edema, pneumothorax or sedative overdose
* No SpO2 signal
* Encephalopathy score > 2
* Delirium
* Other respiratory support needed (intubation or NIV)
* Patient on withdrawal life support
* Advance neoplasia (palliative stage) or terminal respiratory distress
* Unavailability of FreeO2 device at the randomisation
* Non optimal patient collaboration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
Hospital length of stay | From hospital admission until hospital discharge (around one week expected)
  Duration of the hospital length of stay

SECONDARY OUTCOMES:
ICU transfer | During hospital stay : from hospital admission until hospital discharge (around one week expected)
  The rate of ICU admission during hospital stay
Oxygen administration duration | During hospital stay : from hospital admission until hospital discharge (around one week expected)
  The number of days patient receive oxygen supplementation
Non invasive or invasive mechanic ventilation rate use | During hospital stay: from hospital admission until hospital discharge (around one week expected)
  The rate of NIV use during length of stay in hospital

OTHER OUTCOMES:
Arterial or Capillary blood gaz evolution | During hospital stay - From hospital admission until hospital discharge (around one week expected)
  Evaluation of the rate of respiratory acidosis (pH<7.35 and PaCO2>45mmHg)
Hospital Readmission rate after hospital discharge | Until day 90 after study inclusion
  Rate of hospital readmission after initial hospital discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No